CLINICAL TRIAL: NCT03118284
Title: Foley Catheter Related Bladder Discomfort (FCRBD): Role of Neutrophil Cells
Acronym: FCRBD
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator is leaving university and halting studies
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201609072
Record Dates: First submitted 2017-04-05; First posted 2017-04-18 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Urethra Injury; Catheter Site Discomfort
Keywords: Foley catheter
MeSH Terms: interventions — Urine Specimen Collection; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — mtDNA samples isolated from blood and supernatants from urine will be retained and frozen for future research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Foley catheter group: Urine collection and blood collection and NRS for pain in patients having surgery for which their surgeon has ordered placement of a Foley catheter.
  Interventions: Other: urine collection; Other: Blood collection; Behavioral: NRS
- Healthy control group: Blood collection in healthy volunteers from the Research Participant Registry or recruited from posters around the Washington University campus
  Interventions: Other: Blood collection

INTERVENTIONS:
Other: urine collection
  Groups: Foley catheter group
Other: Blood collection
Behavioral: NRS
  Groups: Foley catheter group

SUMMARY:
Urinary [Foley] catheters [tubes] are commonly placed in patients undergoing surgery; approximately 25% of surgical patients will receive one. Among patients who receive urinary catheters, discomfort associated with the Foley catheter is common; between 47-90% of patients experience catheter related bladder discomfort [CRBD]. Presence of a foreign object in the bladder even for short periods of time may result in symptoms such as a burning sensation, pain in the lower abdomen, muscle spasms and a sense of urgency to urinate. There is some evidence that suggests that hospital-acquired urinary tract infections are directly related to catheter placement, which causes mechanical damage and local inflammation to the urethra and the bladder. Based on research conducted on a similar mechanism where an airway tube is inserted into a patients throat for delivery of general anesthesia - we hypothesize that CRBD is related to injury and inflammation caused by the catheter placement and that this occurs in a sterile environment.

DETAILED DESCRIPTION:
Urinary catheterization has been implicated in up to 80% of hospital-acquired UTIs, and has been associated with evidence for immunological and histological damage frequently in the absence of bacteria31. In a recent human study in elderly patients with ASB and UTI analysis of neutrophil activity showed evidence of enzymatic involvement during bladder infection32, and some appeared to relate to pain and inflammation, however no analysis was conducted regarding neutrophil phenotypes and the impact of mtDNA on sterile local injury mediated exclusively by a Foley catheter.

The bladder irritation that results from Foley catheterization appears to be mediated by muscarinic receptors that mediate involuntary bladder smooth-muscle contractility. Thus the main therapy relies on agents with anti-muscarinic activity such as oxybutynin, tolterodine and butylscopolamine, whereas some benefit has been shown with tramadol, ketamine, paracetamol, pregabalin and gabapentin. However no single commonly accepted therapy for FCRBD is available, and there is uncertainty about the safety and efficacy of the current treatments available. Some research has suggested a role for inflammatory mediators in the occurrence of FCRBD as evident by induction of prostaglandin synthesis and cyclooxygenase-2 (COX-2) inhibitors alleviating symptoms related to FCRBD. In summary various therapies to control FCRBD are available but none have directly addressed the acute inflammatory reaction likely mediating these symptoms1,2,3,4. Hence our interest in analyzing the activity of acute inflammatory cells in particular neutrophil activation as a mediator of bladder inflammation and trigger of FCRBD.

Although the exact pathophysiology of FCRBD has not been elucidated, we recently showed expression of inflammatory mediators, neutrophil infiltration and mucosal surface injury in the absence of bacterial infection using a human model of tracheal injury. As it has been clearly shown that neutrophil infiltration and activation can be driven in response to sterile cell death8, our preliminary data suggest that the link between Foley catheter and possible bladder neutrophil accumulation is through mucosal cell injury.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 to 75.
2. American Society of Anesthesiologists Physical Status Classification (ASA) I, II, and III, per CPAP assessment.
3. Planned Foley catheter placement with surgery and hospitalization.
4. Scheduled elective surgery (i.e., orthopedic, neurosurgical, spine surgery, cardiac, thoracic surgery, ear nose and throat surgery).
5. Anticipated length of Foley catheter requirement up to 72 hours.
6. Ability to provide informed consent.

Exclusion Criteria:

1. Visible blood in the urine as evident upon sample collection.
2. More than one attempt to place the Foley catheter as documented by RN in OR.
3. Planned surgical procedure involving the urinary system
4. On dialysis and/or anuric
5. Urinary tract infection (UTI) as documented by primary team within 24 hours of surgery
6. Pregnancy or lactating.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having elective surgery requiring hospitalization and Foley catheter placement.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2017-08-21 (Actual); Study Completion 2017-08-28 (Actual)

PRIMARY OUTCOMES:
Neutrophil surface marker changes in subjects that experience Foley catheter related bladder discomfort [FCRBD] | Change from baseline [immediately after catheter placement] until catheter removal [post-operative day 1, 2, 3].
  Changes in surface inflammatory markers on polymorphonuclear neutrophils associated with bladder injury secondary to Foley catheter placement.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No